CLINICAL TRIAL: NCT05150626
Title: An Open-label, Randomized, Three-period, Crossover, Single-dose Study to Evaluate the Effect of a Low-fat Meal and a Standard Meal on the Pharmacokinetics of DBPR108 in Healthy Subjects
Brief Title: A Study to Evaluate the Effect of Different Meal Types on the Pharmacokinetics of DBPR108 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HA1118-013
Record Dates: First submitted 2021-11-26; First posted 2021-12-09 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — DBPR108

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sequence A administered DBPR108 (Experimental): Subjects will receive a single dose of DBPR108 100 mg under fasted condition, following a low-fat meal and a standard meal.
  Interventions: Drug: DBPR108 tablets
- Sequence B administered DBPR108 (Experimental): Subjects will receive a single dose of DBPR108 100 mg following a low-fat meal and standard meal, under fasted condition.
  Interventions: Drug: DBPR108 tablets
- Sequence C administered DBPR108 (Experimental): Subjects will receive a single dose of DBPR108 100 mg following a standard meal, under fasted condition, following a low-fat meal.
  Interventions: Drug: DBPR108 tablets

INTERVENTIONS:
Drug: DBPR108 tablets — Drug: DBPR108, tablets, oral

SUMMARY:
This is an open-label, randomized, three-period, crossover, single-dose study to evaluate the effects of a low-fat meal and a standard meal on the pharmacokinetics of DBPR108 and the safety and tolerability of DBPR108 under different fed states in healthy adult subjects.

DETAILED DESCRIPTION:
The objective of the study is to evaluate the effect of different meal types on the pharmacokinetics of DBPR108, a potent dipeptidylpeptidase-4 inhibitor. In this open-label, randomized, three-period, crossover study, healthy subjects will receive a single dose of DBPR108 100 mg under fasted conditions and following a low-fat meal or a standard meal. Twenty-one healthy subjects will be randomized 1:1:1 to Sequence A, Sequence B, or Sequence C. This study will consist of a screening and baseline period, a treatment period, and a follow-up period. Blood samples for pharmacokinetic assessments will be taken pre-dose and up to 48 h post-dose.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects fully understand and voluntarily participate in this study and sign informed consent;
2. Healthy male and/or female subjects between the ages of 18 and 45 years (inclusive);
3. Body Mass Index (BMI) of 18 to 28 kg/m2 (inclusive), body weight for male ≥50.0 kg and for female≥45.0 kg；
4. Subjects (including their partners) are willing to use effective contraceptives from screening to the 6 months after the last dose administration;
5. Subjects judged to be in good health by the investigator, based on the physical examination, vital signs examination, 12-lead electrocardiogram (ECG) examination and laboratory examination etc;

Exclusion Criteria:

1. History of allergic conditions, or allergic to any ingredients of DBPR108;
2. History of severe diseases, such as cardiovascular, respiratory, liver, gastrointestinal, endocrine, hematological, psychiatric/neurological systems diseases within 1 year prior to screening;
3. History of hypoglycemia or abnormal blood glucose at screening: fasting blood glucose <70 mg/dL (3.9 mmol/L) or >110 mg/dL (6.1 mmol/L);
4. Subjects who have previously undergone surgery (e.g., subtotal gastrectomy) that may affect the absorption, distribution, metabolism, or excretion of the drug, or who have a scheduled surgery during the study period;
5. History of drug abuse, or urine drug screening is positive at screening;
6. Smoking more than 5 cigarettes per day within 3 months prior to screening, or who cannot stop using nicotine-containing products during the study period;
7. Regular alcohol consumption exceeding 15 g/day(female) or 25 g/day(male) (15 g ≈ 450 mL beer, or 50 mL hard liquor, or 150 mL wine) within the 3 months prior to screening, or taking any product containing alcohol within 48 h before dosing, or alcohol test is positive;
8. Blood donation (or blood loss) ≥400 mL, or receiving blood product transfusion within 3 months prior to screening;
9. Consumption of grapefruit juice, methylxanthine-rich food or beverage (such as coffee, tea, cola, chocolate, energy drinks), or those who have had strenuous exercise, or have other factors affecting drug absorption, distribution, metabolism, excretion, within 48 h before the administration;
10. Use of any prescription drug, over-the-counter drug (except acetaminophen and some nasal sprays), or herbal medicine within 2 weeks prior to screening;
11. Have special dietary requirements and cannot consume the study meals;
12. Subject with hepatitis B surface antigen, hepatitis C virus antibody, human immunodeficiency virus antibody or Treponema pallidum antibody positive;
13. Enrolled in any other clinical trial within 3 months before screening (whichever is administrated);
14. Have been vaccinated within 4 weeks prior to screening or who have a scheduled vaccination during the study period;
15. Pregnant/lactating woman, or who has a positive blood pregnancy test at screening;
16. Not suitable for this study as decided by the investigator due to other reasons.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2022-05-29 (Actual); Primary Completion 2022-06-07 (Actual); Study Completion 2022-07-14 (Actual)

PRIMARY OUTCOMES:
Peak plasma concentration (Cmax) of DBPR108 | Predose and at prespecified time point after DBPR108 dosing on Day 1, Day 5 and Day 9.
Area under the plasma concentration versus time curve from time zero to the time of last measurable concentration (AUClast) of DBPR108 | Predose and at prespecified time point after DBPR108 dosing on Day 1, Day 5 and Day 9.
Area under the plasma concentration versus time curve from time zero to infinity (AUCinf) of DBPR108 | Predose and at prespecified time point after DBPR108 dosing on Day 1, Day 5 and Day 9.

SECONDARY OUTCOMES:
Time to achieve maximum plasma concentration (Tmax) of DBPR108 | Predose and at prespecified time point after DBPR108 dosing on Day 1, Day 5 and Day 9.
Half-life (t1/2) of DBPR108 | Predose and at prespecified time point after DBPR108 dosing on Day 1, Day 5 and Day 9.
Apparent clearance (CL/F) of DBPR108 | Predose and at prespecified time point after DBPR108 dosing on Day 1, Day 5 and Day 9.
Apparent volume of Distribution (Vz/F) of DBPR108 | Predose and at prespecified time point after DBPR108 dosing on Day 1, Day 5 and Day 9.
Number of subjects with treatment-related adverse events as assessed by CTCAE v5.0 | Day 1 to Day 14

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of Soochow University, Suzhou, China